CLINICAL TRIAL: NCT05304559
Title: Effects of S-ketamine and Continuous Iliac Fascia Space Block on Perioperative Neurological Cognitive Impairment and Postoperative Rehabilitation in Elderly Patients With Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Yangtian Shuang, Resident physician, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YShuang
Record Dates: First submitted 2022-03-01; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hip Fractures
Keywords: cognitive dysfunction; s-ketamine; nerve block
MeSH Terms: conditions — Hip Fractures; Cognitive Dysfunction | interventions — Esketamine; Control Groups; Saline Solution

STUDY DESIGN:
Intervention Model Description: A total of 108 patients were enrolled in this trial (the control group was shared by the two schemes). Research drug (esmolamine) test group: control group was designed at 1:1, 36 cases in each group. Research technique (continuous iliac fascia space block) test group: control group was designed at 1:1, 36 cases in each group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug group (Experimental): S-ketamine 0.1mg/kg was injected intravenously during anesthesia induction and esmolamine 0.1mg/ (kg.h) was injected intravenously during anesthesia maintenance.S-Ketamine was put into the analgesia pump as an adjuvant for continuous analgesia until 2 days after operation.
  Interventions: Drug: S-Ketamine
- Device group (Experimental): The hip fracture was diagnosed clinically on admission and ultrasound-guided iliofascial space block was performed after evaluation, and the analgesia lasted until 2 days after operation.
  Interventions: Device: Continuous iliac fascia space block
- Normal saline group (Placebo Comparator): normal saline 0.1ml/kg was injected intravenously during anesthesia induction and normal saline 0.1ml/ (kg.h) was injected intravenously during anesthesia maintenance.normal saline was put into the analgesia pump as an adjuvant for continuous analgesia until 2 days after operation.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: S-Ketamine — S-Ketamine0.1mg/kg was injected intravenously during anesthesia induction and S-Ketamine0.1mg/ (kg.h) was injected intravenously during anesthesia maintenance.S-Ketamine was put into the analgesia pump as an adjuvant for continuous analgesia until 2 days after operation.
  Other Names: control group
  Arms: Drug group
Device: Continuous iliac fascia space block — After admission, the iliac fascia space block and catheterization were performed under the guidance of ultrasound, and the analgesia was continued until two days after operation.
  Other Names: control group
  Arms: Device group
Drug: Normal saline — Normal saline0.1ml/kg was injected intravenously during anesthesia induction and Normal saline0.1ml/ (kg.h) was injected intravenously during anesthesia maintenance.Normal saline was put into the analgesia pump as an adjuvant for continuous analgesia until 2 days after operation.
  Arms: Normal saline group

SUMMARY:
Elderly patients with hip fracture are older and have a high incidence of perioperative complications. the postoperative recovery of elderly patients with hip fracture is affected by hemodynamic instability and pain caused by fracture. S-ketamine is the S-isomer of ketamine. Compared with traditional ketamine, S-ketamine has stronger analgesic effect and fewer adverse reactions of nervous system. The parasympathetic effect of S-ketamine can antagonize the circulatory inhibition of propofol and make the hemodynamics more stable in elderly patients with hip fracture.Iliac fascial space block (fasciailiacacompartmentblock,FICB) mainly depends on local anesthetics spreading to the femoral nerve, lateral femoral cutaneous nerve and obturator nerve in the iliofascial space to achieve analgesia in its dominant area. Ultrasound-guided iliac fascial space block can effectively reduce the amount of anesthetics and has shorter puncture time and fewer complications. It can more effectively reduce the perioperative pain of elderly patients with hip fracture.

DETAILED DESCRIPTION:
With the advent of the aging society, the incidence of hip fracture in elderly patients is increasing year by year, and the incidence of perioperative neurological cognitive impairment (PND) is increasing year by year. PND refers to postoperative brain dysfunction in patients without mental disorders, including postoperative delirium POD and postoperative cognitive dysfunction POCD. PND is more common in clinic, especially in the elderly. The main feature of PND is the long-term decline and decline of cognitive function after operation. PND not only prolongs the length of stay of patients, interferes with postoperative treatment, but even increases mortality. The pathogenesis of PND is not clear, and it is affected by many factors. Studies have shown that keeping intraoperative blood pressure at baseline to 10% above baseline can significantly reduce the incidence of PND. In addition, pain is also an important factor leading to the occurrence of PND. S-ketamine is the S-isomer of ketamine. Compared with traditional ketamine, S-ketamine has stronger analgesic effect and fewer adverse reactions of nervous system. The parasympathetic effect of S-ketamine can antagonize the circulatory inhibition of propofol and make the hemodynamics more stable. Iliac fascial space block (fasciailiacacompartmentblock,FICB) mainly depends on local anesthetics spreading to the femoral nerve, lateral femoral cutaneous nerve and obturator nerve in the iliofascial space to achieve analgesia in its dominant area. Ultrasound-guided iliac fascial space block can effectively reduce the amount of anesthetics and has shorter puncture time and fewer complications. In this study, a randomized controlled trial was conducted to observe the clinical effects of S-ketamine and ultrasound-guided iliac fascia block combined with general anesthesia in elderly patients with hip fracture, and to evaluate their clinical value.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of hip fracture

Aged 65 or above

ASA Ⅰ-Ⅲ

No mental and nervous system diseases

No pathological fractures, such as bone tumor, bone tuberculosis, osteomyelitis, etc

No puncture site infection

No hospital stay for more than 48 hours after operation

Exclusion Criteria:

Patients with severe cardiac, hepatic and renal dysfunction before operation

Long-term use of analgesics, sedatives and alcoholism

Patients with respiratory tract management difficulties (modified Ma's score is IV)

Previous neuropsychiatric diseases such as severe cerebrovascular, Alzheimer's disease, epilepsy and Parkinson's disease

Previous history of intracranial surgery or craniocerebral injury

Severe vision, hearing, language impairment or other reasons unable to communicate

Allergic or contraindicated to ropivacaine or non-steroidal anti-inflammatory drugs (NSAID)

Emergency surgery or trauma patients.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-03-26 (Estimated); Primary Completion 2022-04-26 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
incidence of peioperative neurocognitive impairment | Perioperative period
  incidence of peioperative neurocognitive impairment

CONTACTS AND LOCATIONS:
Overall Officials: jJianhong Sun, master, Study Chair — Yangzhou University
Locations (1):
- Affiliated Hospital of Yangzhou University, Yangzhou, China